CLINICAL TRIAL: NCT04687293
Title: Investigation of the Effectiveness of Rehabilitation Using the HUBER 360 Tool to Reduce the Risk of Falls in People in Pathological Situations Requiring Functional Rehabilitation
Brief Title: Rehabiliation Using HUBER 360 to Reduce the Risk of Falls
Acronym: HUBER-FALLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Charlotte Beaudart, Principal investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUBER_CNRF01
Record Dates: First submitted 2020-12-09; First posted 2020-12-29 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Rehabilitation; Exercise Therapy; Treatment Outcome; Quality of Life; Fall
Keywords: Huber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUBER (Experimental): HUBER is an isometric strengthening device. It consists of an oval motorized platform, which performs rotating, oscillatory movements with a controlled amplitude and speed.
  Intervention will consist of 2 sessions of HUBER per week. Each session lasts approximatively 30 minutes. The intervention is 8 weeks long.
  Interventions: Device: HUBER (LPG Systems, France)
- Control (No Intervention): The control group will not received any intervention except usual care.

INTERVENTIONS:
Device: HUBER (LPG Systems, France) — The HUBER® device consists of an oval motorized platform, which performs rotating, oscillatory movements with a controlled amplitude and speed. It also comprises, two large handles with force sensors, mounted on a movable column. Its originality is based on its capacity to capture simultaneously the subjects' balance, core stability, core strength and total body strength; and adapt the training accordingly. Indeed, the platform interferes with the balance of the patient who must continually adjust his/her posture by exerting isometric pushing and pulling efforts with the arms. As a result, the device provides postural and muscle adaptation with visual feedback. Due to the constant adaptation of the device, it is thought to enhance muscular strength and improve neuromuscular coordination simultaneously.
  Arms: HUBER

SUMMARY:
Aim: The aim of the present study was to analyse the effects of training performed on a rotating, motorised platform (the Huber/SpineForce device from LPG Systems, Valence, France) intended to reduce the risk of falls.

Subjects: any patient 1) benefiting from a physiotherapy rehabilitation program at the CHU Liège, CNRF, Belgium; 2) presenting a pathological situation justifying functional rehabilitation with HUBER 360®; 3) presenting any pathology not constituting an exclusion criterion; 4) giving informed consent to research will be include in this 8-week interventional trial.

Design: randomized open-label trial. Patients will be randomized into the intervention group (HUBER trainig, 45 minutes of training, twice a week during 8 weeks) or in the control group (standard care).

Outcomes: the effect of the training will be measured on the Time-Up-and-Go test, on the Short-Physical performance battery test and on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient benefiting from a physiotherapy rehabilitation program at the CHU Liège, CNRF
* Patient presenting a pathological situation justifying functional rehabilitation with HUBER 360®
* Patient presenting any pathology not constituting an exclusion criterion
* Patient giving informed consent to research.

Exclusion Criteria:

* Cardiac or respiratory or neurological or rheumatological disease incompatible with physical activity ;
* Joint inflammation;
* Rheumatic disease in acute phase;
* Recent trauma, infection of the musculoskeletal system;
* Fever;
* Venous thrombosis ;
* Discopathy in acute phase;
* Neuropsychological problems that do not allow to integrate the instructions or other serious psychological problems;
* Cardiovascular diseases and any progressive, chronic, counter-indicative disease;
* Large anatomical deformities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Risk of falls, in seconds | 8 weeks
  Measured with Timed-Up-and Go test

SECONDARY OUTCOMES:
Physical performance | 8 weeks
  Short Physical Performance Battery test (SPPB test). The test is scored from 0 (lower physical performance) to 12 (highest physical performance)
Quality of life, measured with the Short Form-36 questionnaire | 8 weeks
  SF-36 generic quality of life questionnaire. The score obtained from this questionnaire is composed with a Physcial component Scale (PMS) and a Mental component scale (MCS). Results are scored from 0 (worst quality of life) to 100 (best quality of life).
Utility score using the EuroQol- 5 Dimension questionnaire | 8 weeks
  Descriptive data from the 5 dimensions can be used to generate a health-related quality of life profile for the subject. The questionnaire is scored from 0 (worst health state imaginable) to 100 (best health state imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Kaux, MD PhD, Study Director — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU Liège, CNRF, Tinlot, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No